CLINICAL TRIAL: NCT06749743
Title: Accuracy Of Dental Caries Detection From Intraoral Images Using Different Artificial Intelligence Models Versus Conventional Visual Examination Among A Group Of Children: A Diagnostic Accuracy Study
Brief Title: Accuracy Of Detection Of Dental Caries From Intraoral Images Using Different ArtificiaI Intelligence Models
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherine Tarek Mohamed Elsayed Khaled, principal investigator, Cairo University
Other Study IDs: OP 7-1-1
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries (Diagnosis); Artifical Intelligence; Intraoral Images
Keywords: artificial intelligence; dental caries; diagnosis; intraoral images
MeSH Terms: conditions — Dental Caries; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- training group: images used to train the AI models on detection of dental caries from intraoral images.
  Interventions: Diagnostic Test: FASTER RCNN
- test group: images used to test the accuracy of the AI models in diagnosis of dental caries from intraoral images.
  Interventions: Diagnostic Test: FASTER RCNN

INTERVENTIONS:
Diagnostic Test: FASTER RCNN — train artificial intelligence models ( FASTER RCNN, YOLOY ) to detect dental caries , then test their accuracy
  Other Names: YOLO

SUMMARY:
The goal of this observational study is to evaluate the diagnostic accuracy of different deep learning models in detecting dental caries from intra oral images taken by a professional intra oral camera in children. The main question it aims to answer is:

What is the diagnostic accuracy of different deep learning models in detecting dental caries from intra oral images taken by a professional intra oral camera in children compared to the conventional clinical visual examination?

ELIGIBILITY:
Inclusion Criteria:

* Child dentition having at least one decayed tooth.

Exclusion Criteria:

* Child dentition with developmental enamel defects.
* Children with any systemic medical condition.
* Parent / child refuse to participate in the study.
* Uncooperative child.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child with at least one decayed tooth present at the time of recruitment at the Pediatric dental department diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy Of Dental Caries Detection From Intraoral Images Using Different Artificial Intelligence Models Versus Conventional Visual Examination Among A Group Of Children: A Diagnostic Accuracy Study | one year
  Diagnostic accuracy of index tests will be determined, including sensitivity, specificity, overall accuracy, positive and negative predictive values and ROC curve analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided